CLINICAL TRIAL: NCT02729324
Title: Comparison of Efficacy and Safety Between Medical Radiation Protectants (FORRAD®) and Trolamine (Biafine) for the Management of Radiation Dermatitis in Patients With Nasopharyngeal Carcinoma Receiving IMRT: A Single-center, Randomized Controlled Trial
Brief Title: Comparison of Efficacy and Safety Between Medical Radiation Protectants (FORRAD®) and Trolamine (Biafine) for the Management of Radiation Dermatitis in Patients With Nasopharyngeal Carcinoma Receiving IMRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yun-fei Xia (Other)
Responsible Party: Sponsor-Investigator, Yun-fei Xia, Director of Department of Radiation Oncology, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B2015-071-01
Record Dates: First submitted 2016-03-27; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Nasopharyngeal Neoplasms; Radiodermatitis
Keywords: nasopharyngeal carcinoma (NPC); radiation dermatitis; intensity modulated radiation therapy (IMRT)
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Radiodermatitis; Nasopharyngeal Carcinoma | interventions — triethanolamine; Biafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FORRAD group (Experimental): This group of patients will receive Medical Radiation Protectants (FORRAD®) during study for prevention and treatment of acute radiation-induced dermatitis. This is the experimental group.
  Interventions: Drug: Medical Radiation Protectants (FORRAD®)
- Biafine group (Active Comparator): This group of patients will receive Trolamine (Biafine) during study for prevention and treatment of acute radiation-induced dermatitis. This is the active comparator group.
  Interventions: Drug: Trolamine (Biafine)

INTERVENTIONS:
Drug: Medical Radiation Protectants (FORRAD®) — Medical Radiation Protectants (FORRAD®) is prescribed at the beginning of radiotherapy for free. Patients are asked to start topical application of Medical Radiation Protectants (FORRAD®) on irradiated skin at the onset of radiotherapy, three times a day (30 minutes before radiotherapy, after radiotherapy, and before bedtime), until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation dermatitis. When grade 2 or higher radiation dermatitis is developed, patients can continue using Medical Radiation Protectants (FORRAD®). When grade 3 or higher radiation dermatitis happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted, until moist desquamation is cured.
  Arms: FORRAD group
Drug: Trolamine (Biafine) — Trolamine (Biafine) is prescribed at the beginning of radiotherapy. Patients are asked to start topical application of trolamine (Biafine) on irradiated skin at the onset of radiotherapy, three times a day, until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation dermatitis. No other prophylactic creams, lotions, or gels are allowed. When grade 2 or higher radiation dermatitis is developed, patients cannot use trolamine any more, and they will receive other conventional medical care for treatment of radiation dermatitis in the investigators institution. When grade 3 or higher radiation dermatitis happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted, until moist desquamation is cured.
  Arms: Biafine group

SUMMARY:
Radiation therapy remains the principal treatment for nasopharyngeal carcinoma (NPC). Although intensity modulated radiation therapy (IMRT) has been widely used in China nowadays, radiation dermatitis is still common. It has an impact on pain and quality of life, and if severe, may lead to interruption of the radiation schedule for the patient. Trolamine (Biafine; Genmedix Ltd, France) is commonly prescribed at the beginning of radiotherapy for preventing acute radiation-induced skin toxicity in China. However, as long as grade ≥2 radiation dermatitis is developed, trolamine is not allowed to use any more. Medical Radiation Protectants (FORRAD®) is a new kind of topical agents for prevention and treatment of radiation dermatitis. It could be used during the course of radiotherapy, even when grade ≥2 dermatitis is developed. This randomized phase II study is aimed to assess the effectiveness and safety of Medical Radiation Protectants (FORRAD®) for the prevention and treatment of acute radiation-induced dermatitis of grade 3 or higher during IMRT for patients with NPC, compared with trolamine.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignances in South China. Radiation therapy remains the principal treatment for NPC. One of the frequently occurred radiation-related side effects includes radiation-induced skin reactions (RISR), also known as radiation dermatitis, which affects up to 90% of cancer patients receiving radiation therapy. Although intensity modulated radiation therapy (IMRT) has been widely used in China nowadays, radiation dermatitis is still common. It is often characterized by edema, erythema, changes in pigmentation, fibrosis, and ulceration, and may cause signs and symptoms, such as skin dryness, itching discomfort, pain, warmth, and burning. Radiation dermatitis has an impact on pain and quality of life in this patient group, and if severe, may lead to interruption of the radiation schedule for the patient.

A variety of interventions are used for prophylaxis and management of radiation dermatitis. However, a recent overview of systematic review and meta-analysis of randomized controlled trials concluded that the use of these interventions is not yet supported by conclusive evidence and therefore warrants further investigations.

Trolamine (Biafine; Genmedix Ltd, France) is an oil-in-water emulsion that can enhance skin healing by recruiting macrophages and modifying the concentrations of various immunomodulators. In China, Trolamine is commonly prescribed at the beginning of radiotherapy for preventing acute radiation-induced skin toxicity. However, as long as grade ≥2 radiation dermatitis is developed, Trolamine is not allowed to use any more. Medical Radiation Protectants (FORRAD®) is a new kind of topical agents for prevention and treatment of radiation dermatitis. It could be used during the course of radiotherapy, even when grade ≥2 dermatitis is developed.

The primary aim of this randomized phase II study is to assess the effectiveness and safety of Medical Radiation Protectants (FORRAD®) for the prevention and treatment of acute radiation-induced dermatitis of grade 3 or higher during IMRT for patients with NPC, compared with trolamine.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed and previously untreated nasopharyngeal carcinoma.
2. Age ≥ 18 years and ≤ 65 years.
3. Karnofsky performance status (KPS) score ≥ 70.
4. No prior radiation or surgery in the head and neck.
5. No contraindication to radiotherapy.
6. Planned to receive radiotherapy alone or concurrent chemoradiotherapy, with intensity-modulated radiation therapy (IMRT).
7. Adequate bone marrow function: while blood cell >= 3,000/μL, absolute neutrophil count >= 1,500/μL, hemoglobin >= 100g/L, platelet >= 75,000/μL.
8. Life expectancy of >= 3 months.

Exclusion Criteria:

1. Known allergic reaction to any component of Medical Radiation Protectants (FORRAD®) or Trolamine (Biafine), or severe allergic constitution.
2. Other conditions that the investigators consider as inappropriate for enrolling into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 radiation dermatitis | Day 56 after completion or termination of radiotherapy
  Incidence of grade ≥ 3 radiation dermatitis according to CTCAE version 4.0
The Skindex-16 | Day 56 after completion or termination of radiotherapy
  The skindex-16 is an analogue scale of symptoms and functional endpoints related to skin toxicity that may occur in the radiation treatment area. The mean AUC of Skindex-16 score over time. Patients were asked to complete the Skindex-16 only in reference to the skin receiving RT.
The symptom experience diary (SED) | Day 56 after completion or termination of radiotherapy
  The symptom experience diary (SED) required the patient to rate the severity of multiple skin toxicity-related signs and symptoms on a scale of 0 (do not experience) to 10 (experience all the time).
EORTC QLQ-C30 | Day 56 after completion or termination of radiotherapy
  EORTC QLQ-C30 is a Quality-of-Life Instrument proposed by the European Organization for Research and Treatment of Cancer (EORTC), for use in International Clinical Trials in Oncology. The QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.

SECONDARY OUTCOMES:
Interruption time during the schedule of radiotherapy | Through radiotherapy completion or termination, an average of 7 weeks
  The cumulative interruption time during the schedule of radiotherapy because of grade 3 or higher radiation dermatitis.
Time for healing of radiation dermatitis | Through study completion, an average of 15 weeks
  Time until healing of radiation dermatitis, after the completion or the termination of radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Zhang LF, Li YH, Xie SH, Ling W, Chen SH, Liu Q, Huang QH, Cao SM. Incidence trend of nasopharyngeal carcinoma from 1987 to 2011 in Sihui County, Guangdong Province, South China: an age-period-cohort analysis. Chin J Cancer. 2015 May 14;34(8):350-7. doi: 10.1186/s40880-015-0018-6. PMID 26058679
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Mao YP, Yin WJ, Guo R, Zhang GS, Fang JL, Chi F, Qi ZY, Liu MZ, Ma J, Sun Y. Dosimetric benefit to organs at risk following margin reductions in nasopharyngeal carcinoma treated with intensity-modulated radiation therapy. Chin J Cancer. 2015 May 20;34(5):189-97. doi: 10.1186/s40880-015-0016-8. PMID 26058563
- [Background] Zheng Y, Han F, Xiao W, Xiang Y, Lu L, Deng X, Cui N, Zhao C. Analysis of late toxicity in nasopharyngeal carcinoma patients treated with intensity modulated radiation therapy. Radiat Oncol. 2015 Jan 13;10:17. doi: 10.1186/s13014-014-0326-z. PMID 25582731
- [Background] Chan RJ, Webster J, Chung B, Marquart L, Ahmed M, Garantziotis S. Prevention and treatment of acute radiation-induced skin reactions: a systematic review and meta-analysis of randomized controlled trials. BMC Cancer. 2014 Jan 31;14:53. doi: 10.1186/1471-2407-14-53. PMID 24484999
- [Background] Elliott EA, Wright JR, Swann RS, Nguyen-Tan F, Takita C, Bucci MK, Garden AS, Kim H, Hug EB, Ryu J, Greenberg M, Saxton JP, Ang K, Berk L; Radiation Therapy Oncology Group Trial 99-13. Phase III Trial of an emulsion containing trolamine for the prevention of radiation dermatitis in patients with advanced squamous cell carcinoma of the head and neck: results of Radiation Therapy Oncology Group Trial 99-13. J Clin Oncol. 2006 May 1;24(13):2092-7. doi: 10.1200/JCO.2005.04.9148. PMID 16648511
- [Background] Rollmann DC, Novotny PJ, Petersen IA, Garces YI, Bauer HJ, Yan ES, Wahner-Roedler D, Vincent A, Sloan JA, Issa Laack NN. Double-Blind, Placebo-Controlled Pilot Study of Processed Ultra Emu Oil Versus Placebo in the Prevention of Radiation Dermatitis. Int J Radiat Oncol Biol Phys. 2015 Jul 1;92(3):650-8. doi: 10.1016/j.ijrobp.2015.02.028. Epub 2015 Apr 28. PMID 25936812
- [Background] Fisher J, Scott C, Stevens R, Marconi B, Champion L, Freedman GM, Asrari F, Pilepich MV, Gagnon JD, Wong G. Randomized phase III study comparing Best Supportive Care to Biafine as a prophylactic agent for radiation-induced skin toxicity for women undergoing breast irradiation: Radiation Therapy Oncology Group (RTOG) 97-13. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1307-10. doi: 10.1016/s0360-3016(00)00782-3. PMID 11121627
- [Background] Pommier P, Gomez F, Sunyach MP, D'Hombres A, Carrie C, Montbarbon X. Phase III randomized trial of Calendula officinalis compared with trolamine for the prevention of acute dermatitis during irradiation for breast cancer. J Clin Oncol. 2004 Apr 15;22(8):1447-53. doi: 10.1200/JCO.2004.07.063. PMID 15084618